CLINICAL TRIAL: NCT03975270
Title: An Exploratory Study of Sintilimab in Combination With Nab-paclitaxel in Patients With Advanced Recurrent or Metastatic HNSCC (Head and Neck Squamous Cell Carcinoma )After 2 or More Prior Lines of Therapy
Brief Title: Sintilimab in Combination With Nab-paclitaxel in Patients With HNSCC (Head and Neck Squamous Cell Carcinoma )
Acronym: HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengyu Zhou (Unknown)
Responsible Party: Sponsor-Investigator, Shengyu Zhou, vice-director, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSCC-2LIOS-001
Record Dates: First submitted 2019-05-21; First posted 2019-06-05 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Squamous Cell Cancer
MeSH Terms: interventions — sintilimab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab in Combination With Nab-paclitaxe (Experimental): Sintilimab 200 mg intravenous drip, first day Nab-paclitaxe120 mg/m2, intravenous drip, first day and eighth day
  Interventions: Drug: Sintilimab and Nab-paclitaxel

INTERVENTIONS:
Drug: Sintilimab and Nab-paclitaxel — Sintilimab in Combination with Nab-paclitaxel in Patients with Advanced Recurrent or Metastatic HNSCC after 2 or More Prior Lines of Therapy
  Other Names: IBI308

SUMMARY:
Clinical studies related to immunotherapy of HNSCC have shown that PD1 monoclonal antibody has better clinical benefits than conventional chemotherapy. This phase II clinical study is a single arm, open, single-center study. The aim of this study is to observe and evaluate the efficacy and safety of Sintilimab combined with paclitaxel-albumin-binding for injection in patients with advanced recurrent and metastatic HNSCC who fail to receive first-line or more treatment. Participation in this study for treatment may benefit patients with advanced recurrence or metastasis of HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age (> 18 years old) and (< 70 years old) are acceptable for both men and women.
2. Understand the steps and contents of the experiment and sign the written informed consent voluntarily;
3. Histopathology was locally recurrent/metastatic squamous cell carcinoma of the head and neck.
4. In the past, at least one line of platinum-containing chemotherapy or combined with EGFR monoclonal antibody targeting therapy failed or relapsed. Definition of treatment failure: progress after chemotherapy or treatment after ecurrence/metastasis; progress within 6 months after concurrent radiotherapy and chemotherapy can be counted as first-line treatment; all treatment changes due to drug intolerance are not counted as treatment failure;
5. Agree to provide archived specimens of tumor tissue or fresh tissue (not necessarily tissue specimens);
6. ECOG score 0-2;
7. Expected survival of more than 3 months;
8. Computed tomography scans erformed within 28 days prior to the study should show that there is at least one clearly measurable tumor lesion in two vertical directions, the shortest diameter of which is greater than or equal to 1.0 cm (according to RESIST 1.1 standard).
9. Systematic chemotherapy and targeted therapy have been completed for at least 2 weeks before the study, and extensive/local palliative radiotherapy has been completed for at least 4 weeks.
10. Before the study, corticosteroids (prednisone > 10 mg/day or equivalent dose) were discontinued for at least two weeks.
11. Major operations requiring general anesthesia must have been completed for at least four weeks before drug use is studied; operations requiring local anesthesia/epidural anesthesia must have been completed for at least two weeks and the patient has recovered; skin biopsy requiring local anesthesia has been completed for at least one hour;
12. Previous antineoplastic biotherapies (cancer vaccines, cytokines or growth factors for tumour control) were completed for at least four weeks before the study.
13. Hemoglobin (> 90 g/L), neutrophils (> 1.0 *109/L) and platelets (> 80 *109/L) are required for routine blood tests (no blood transfusion or use of biological stimulating factors within 14 days prior to detection).
14. Serum creatinine (< 1.5 *ULN) or creatinine clearance (>50 mL/min) (Cockcroft-Gault formula);
15. Total bilirubin < 1.5 *ULN (Gilbert syndrome allows < 5 *ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 *ULN (patients with liver metastasis allow AST and/or ALT < 5 *ULN);
16. Thyroid function indicators: thyroid stimulating hormone (TSH), free thyroxine (FT3/FT4) in the normal range; if TSH is not in the normal range, FT3/FT4 in the normal range can be included in the group;
17. Adverse reactions caused by previous treatments recovered to grade 1 or below before admission (except for grade 2 neurotoxicity caused by alopecia and chemotherapeutic drugs).
18. Women who were confirmed not to be pregnant within 7 days prior to the study were required to agree to take medically approved effective contraceptive measures throughout the trial period and within 6 months after the end of the trial. 19. Patients can follow up on schedule, communicate well with researchers and complete the study in accordance with the research requirements.

    -

Exclusion Criteria:

1. Patients who meet any of the following conditions will not be allowed to enter the study:
2. Patients diagnosed as nasopharyngeal or thyroid cancer;
3. To clarify the infiltration of the central nervous system (CNS), including brain parenchyma, meningeal invasion or spinal cord compression.
4. History of organ transplantation or hematopoietic stem cell transplantation in the past;
5. Patients with other malignant tumors (excluding cured cervical carcinoma in situ or basal cell or squamous cell carcinoma) may not participate in the study unless they have complete remission for at least five years prior to admission and need no other treatment or treatment during the study period;
6. History of active and known autoimmune diseases, including, but not limited to, systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, with the exception of type I diabetes mellitus, hypothyroidism controlled only by hormone replacement therapy, skin diseases without systemic treatment (such as vitiligo, psoriasis), controlled milk Celiac disease, or disease that is not expected to recur without external stimuli.
7. Anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell co-stimulation or checkpoint pathway) have been used before.
8. Uncontrolled hypertension (systolic pressure > 140 mmHg and/or diastolic pressure > 90 mmHg) or pulmonary hypertension or unstable angina pectoris; myocardial infarction or bypass or stent surgery within 6 months prior to administration; a history of chronic heart failure at NYHA grade 3-4; clinically significant valvular disease; severe arrhythmias requiring treatment, including QTc interval males For women (> 450 ms, 470 ms), left ventricular ejection fraction (LVEF) < 50%, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months before administration, etc.
9. Complicated with serious medical diseases, including but not limited to uncontrolled diabetes, active gastrointestinal ulcer, active hemorrhage, etc.
10. Active infections requiring systemic treatment;
11. Past or current patients with active tuberculosis infection;
12. Acquired immunodeficiency syndrome antibody (Anti-HIV) and anti-Treponema pallidum antibody (TP-Ab) were positive; hepatitis C antibody (HCV-Ab) was positive and hepatitis C virus RNA quantification was higher than the upper limit of detection unit normal value; hepatitis B surface antigen (HBV-Ag) was positive and HBV DNA quantification was higher than the upper limit of detection unit normal value;
13. Complications requiring immunosuppressive drugs or systemic treatment at a dose of immunosuppressive drugs (prednisone > 10mg/day or equivalent dose of the same drug) are allowed to inhale or locally use steroids or doses of prednisone > 10mg/day or equivalent doses of the same drug in the absence of active autoimmune diseases.
14. Other research drugs were used within 30 days prior to the start of the study or within 5 half-lives (whichever is short) of other research drugs; or research instruments were used within 30 days prior to the start of the study.
15. To study the use of live or attenuated vaccines within four weeks before medication.
16. Uncontrolled or markedly symptomatic serous effusion such as pleural, abdominal, pelvic and pericardial effusion;
17. Those who have a history of drug abuse or drug abuse upon inquiry;
18. History of interstitial lung disease;
19. Lactating women are unwilling to stop breastfeeding.
20. Allergies to recombinant humanized monoclonal antibodies or any of their excipients are known; a history of severe allergic diseases is known;
21. Patients do not communicate, understand and cooperate enough, or have poor compliance, which can not guarantee that they can carry out according to the requirements of the program.
22. Researchers believe that for various other reasons, it is not appropriate for participants in this clinical trial to withdraw from the study or terminate the treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  Objective mitigation rate assessed by RECIST 1.1 standard

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College; Beijing Key Laboratory of Clinical Study on Anticancer Molecular Targeted Drugs, Beijing, China